CLINICAL TRIAL: NCT02363231
Title: Maximal Inspiratory Pressure at Extubation: Relationship With Mortality
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, BOUCHRA LAMIA, MD, PhD, University Hospital, Rouen
Other Study IDs: 2013-A01157-38
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients under mechanical ventilation

SUMMARY:
The process of weaning from mechanical ventilation was decided after clinical judgment and weaning predictive index. Nevertheless, indexes predicting weaning outcome like Maximal Inspiratory Pressure (MIP) are frequently inaccurate. However the long-term involvement of respiratory muscles in critically ill patients has not been established. The objective of this study was to assess the relationship on MIP at extubation on one-year mortality in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation at least at 24 hours

Exclusion Criteria:

* Delirium
* Cognitive dysfunction
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patient under invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mortality | One year after extubation

SECONDARY OUTCOMES:
Time to mechanical ventilation weaning | During Intensive care unit hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Clement Medrinal, Principal Investigator — Groupe Hospitalier du Havre
Locations (1):
- Le Havre, Jacques Monod Hospital, Montivilliers, France

REFERENCES:
- [Derived] Combret Y, Prieur G, Hilfiker R, Gravier FE, Smondack P, Contal O, Lamia B, Bonnevie T, Medrinal C. The relationship between maximal expiratory pressure values and critical outcomes in mechanically ventilated patients: a post hoc analysis of an observational study. Ann Intensive Care. 2021 Jan 13;11(1):8. doi: 10.1186/s13613-020-00791-4. PMID 33438092
- [Derived] Medrinal C, Prieur G, Combret Y, Quesada AR, Bonnevie T, Gravier FE, Frenoy E, Contal O, Lamia B. Reliability of respiratory pressure measurements in ventilated and non-ventilated patients in ICU: an observational study. Ann Intensive Care. 2018 Jan 30;8(1):14. doi: 10.1186/s13613-018-0362-1. PMID 29380080
- [Derived] Medrinal C, Prieur G, Frenoy E, Robledo Quesada A, Poncet A, Bonnevie T, Gravier FE, Lamia B, Contal O. Respiratory weakness after mechanical ventilation is associated with one-year mortality - a prospective study. Crit Care. 2016 Jul 31;20(1):231. doi: 10.1186/s13054-016-1418-y. PMID 27475524